CLINICAL TRIAL: NCT06017570
Title: Risk Factors for Distal Caries of Second Molars Adjacent to Mesioangular or Horizontal Partially Erupted Mandibular Third Molars, A Cross-Sectional Study
Brief Title: Risk Factors for Distal Caries of Second Molars Adjacent to Mandibular Impacted Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SelcukU003
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Decay, Dental; Impacted Third Molar Tooth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-risk Group (Experimental): Participants with DMFT score: 0 or 1.
  Interventions: Diagnostic Test: Radiologic examination on orthopantomogram; Diagnostic Test: Clinical examination after surgery
- Modarate-risk Group (Experimental): Participants with DMFT score: 2, 3, 4 or 5.
  Interventions: Diagnostic Test: Radiologic examination on orthopantomogram; Diagnostic Test: Clinical examination after surgery
- High-risk Group (Experimental): Participants with DMFT score above 5.
  Interventions: Diagnostic Test: Radiologic examination on orthopantomogram; Diagnostic Test: Clinical examination after surgery

INTERVENTIONS:
Diagnostic Test: Radiologic examination on orthopantomogram — Caries examination on the distal side of the adjacent second molar in the orthopantomogram of patients with an appointment for the extraction of mesioangular or horizontal partially impacted third molars
Diagnostic Test: Clinical examination after surgery — İnspectional caries examination on the distal side of the adjacent second molar after surgery of patients with mesioangular or horizontal partially impacted third molars

SUMMARY:
Distal surfaces of second molars adjacent to wisdom teeth are always at risk for caries and external root resorption. The incidence of caries is high, especially in partially impacted third molars in mesioangular and horizontal positions. In this study, investigators aimed to examine the caries correlation in the distal second molar with the age, gender, side and DMFT scores of the participants.

ELIGIBILITY:
Inclusion Criteria:

* being between 20 and 40 years old
* having a surgery appointment for removal of the partially impacted third molar which is mesioangular or horizontal position
* having an orthopantomogram on the database
* and having a second molar adjacent to the impacted third molar

Exclusion Criteria:

* crowned or restored the second molar
* any surgery related to the contact area
* any pathology related to the second or third molar
* a radiological artifact on the contact area
* insufficient radiological quality for the evaluation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 639 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Radiologic examination | 10 minute before the start of surgery
  Radiologic examination on the distal side of the second molar for tooth decay
Intra-oral examination | 10 minute before the start of surgery
  Obtaining DMFT score
Clinical examination | 1 minutes after the removal of third molar
  Clinical examination (intra-oral) on the distal side of the second molar for tooth decay

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Gürses, Study Chair — Selcuk University, Faculty of Dentistry
Locations (1):
- Selcuk University, Faculty of Dentistry, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided